CLINICAL TRIAL: NCT02512601
Title: Prospective Evaluation of the Quality of Life of Patients With Post-thrombotic Syndrome Who Receive Compression Therapy and Sulodexide - SQUARES Study
Brief Title: Prospective Evaluation of the QoL of Patients With PTS Who Receive Compression Therapy and Sulodexide
Acronym: SQUARES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor inclusion
Sponsor: Bama GeVe, S.L.U. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SULODEXIDE_PTS/01/13
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Post-thrombotic Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sulodexide (Experimental): Compression therapy + Sulodexide (two capsules of Sulodexide 15 mg twice daily).
  Interventions: Drug: Sulodexide; Other: Compression therapy

INTERVENTIONS:
Drug: Sulodexide — Sulodexide (two capsules of Sulodexide 15 mg twice daily).
  Other Names: Aterina
Other: Compression therapy — Compression:
  * With an orthosis: Compression 22-29 mmHg, length of 20 cm above the DVT area.
  * With a bandage: 7-10 m long and 10 cm wide.
  * Both strategies (orthosis vs bandage) are equally applicable.

SUMMARY:
This study aims to evaluate whether, in a standardised cohort of patients with mild to moderate PTS, monitored for a sufficiently long follow-up period, quality of life measured by generic instruments and disease-specific instruments evolves favourably in this patient profile.

Study objective: to evaluate the evolution of quality of life in general and in the specific context of the disease of patients who have experienced an episode of deep-vein thrombosis (DVT), are affected by post-thrombotic syndrome, are subject to compression therapy and receive an additional standard venoactive agent (sulodexide 15 mg twice daily during 6 months).

DETAILED DESCRIPTION:
Chronic venous insufficiency, or chronic venous disease (CVD), after prior deep-vein thrombosis (DVT), is diagnosed as post-thrombotic syndrome (PTS). It has been calculated that PTS occurs in between 20% and 50% of patients after an episode of DVT, even after having received optimal anticoagulant treatment, and this disorder usually consolidates in the first 2 years after the acute thrombotic episode. The presentation of PTS varies from mild symptoms or clinical signs to severe presentations in approximately 10% of cases, including chronic pain in the limbs that limits activity and ability to work, untreatable oedema and ulcers in the legs.

The cornerstone of the treatment of consolidated PTS is compression treatment, especially in the form of elastic compression stockings, and frequent elevation of the leg, despite the low level of evidence, but these measures require the strictest possible therapeutic compliance on the part of the patient. There is still little evidence that "venoactive" agents are effective in PTS symptoms; nevertheless, the use of medications in PTS is very widespread. In a study by González- Fajardo et al., the use of compression stockings is described in 75% of patients and, in a study by Lozano -Sánchez et al., their use is described in 62% of patients. In the latter study, venoactive drugs were used in approximately 90% of patients.

The diagnosis, staging, prognosis and evolution of the severity of the various entities grouped together under the heading of CVD, including PTS, are based mainly on scales and scoring systems. Objective evaluation of CVD severity tends to be based on the "clinical, etiologic, anatomic and pathophysiologic" (CEAP) clinical classification, the Venous Clinical Severity Score (VCSS) and the Villalta score. Nevertheless, at the present time it is recognised that the assessment of severity does not necessarily coincide with the perception that patients themselves have of their quality of life, which is estimated with generic questionnaires (such as the abbreviated 36-item Short-Form Health Survey questionnaire Short Form (SF-36) and disease-specific questionnaires (such as the Venous Insufficiency Epidemiological and Economic Study questionnaire (VEINES-QOL).

Various studies used some of these scales, usually more than one. All the studies agree that patients with PTS have a lower QoL than those without PTS, and this is shown by both generic and specific instruments. Nonetheless, the population examined in the studies was extremely heterogeneous with respect to use of compression treatment, use of drugs and duration of observations.

The problem that remains to be solved is whether the therapeutic measures applied lead to a change in the QoL measured by generic and disease-specific instruments over a relatively long treatment period. Achieving favourable changes in patients' perception of quality of life remains fundamental for therapeutic compliance and for a suitable physician-patient relationship in the treatment of any chronic disease, and therefore in PTS. This matter can be properly examined, first, in a cohort of patients that is as standardised as possible with respect to the stage and seriousness of the disease and the use of compression treatment and pharmacological treatment.

The standardisation of the stage and seriousness of the disease, as well as the means of standardising the compression treatment, can be achieved with appropriate inclusion and exclusion criteria. As pharmacological treatment is generally administered, sulodexide was chosen for purposes of standardisation. This is a venoactive treatment with antithrombotic, profibrinolytic and endothelium-protective activity, already being used in PTS patients with favourable results. The guidelines of the Society for Vascular Surgery, the American Venous Forum and the American College of Chest Physicians (ACCP) include it among the recommended pharmacological treatments, along with compression, for patients with manifest chronic venous disease. Standardisation of the determination of QoL is envisaged using the generic questionnaire SF-36 and the disease-specific questionnaire VEINES-QOL.

In this way, this study aims to evaluate whether, in a standardised cohort of patients with mild to moderate PTS, monitored for a sufficiently long follow-up period, quality of life measured by generic instruments and disease-specific instruments evolves favourably in this patient profile. If this is the case, a different approach to the treatment of the disease will be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years, ≤ 75 years, of both genders and any ethnic group.
* Prior DVT documented by duplex colour Doppler ultrasound of the lower limbs (if the value of the D dimer and Doppler ultrasound are available, keep them as clinical documentation and note this in the CRF).The previous medical report that documented the prior DVT must be stored in the medical records.
* Post-thrombotic syndrome (PTS) confirmed by duplex colour Doppler ultrasound of the lower limbs.2
* Villalta score ≥ 5. To confirm the presence of PTS at V1, the patient must have a Villalta score ≥ 5 and a positive duplex colour Doppler ultrasound scan of the lower limbs.
* Patients who use compression therapy in accordance with the study requirements. If the patient does not use compression therapy, it must be prescribed at the screening visit (V1) and continued throughout the patient's participation in the study.

During the study, compression therapy must be followed, and compliance will be recorded by the investigator. All patients must have the same degree of compression:

With an orthosis: Compression 22-29 mmHg, length of 20 cm above the DVT area. With a bandage: 7-10 m long and 10 cm wide. Both strategies (orthosis vs bandage) are equally applicable.

* Patients of CEAP class: C0s - C5.
* DVT occurred at least 6 months ago and no more than 5 years ago.
* VEINES-QOL score ≤ 45 at the enrolment visit (V2). For definitive enrolment in the study at the enrolment visit (V2), the patient must have a total score on the VEINES-QOL questionnaire of:

  * Score ≤ 60 adding together the responses to the questions: 1.1-1.9; 4a-4d; 5a-5d; 8a-8e and at the same time
  * Score≥9 adding together the responses: 3; 6; 7 which, after standardisation of the questionnaire responses, must add up to a total VEINES-QOL score ≤ 45.
* Patients with BMI ≤ 40.
* Ability to complete the quality-of-life (QoL) questionnaire.
* Patients able to use the study drug properly.
* Ability to grant informed consent.
* Women of child-bearing age must show a negative result on the urine pregnancy test and use a suitable contraceptive method (not including hormonal contraceptives) throughout the entire period of the study.
* Any possible concomitant treatment with haemorheological, phlebostatic or other venoactive medications must be suspended at the screening visit.

Exclusion Criteria:

* Patients < 18 years or > 75 years.
* BMI > 40.
* Ankle brachial index (ABI) < 0.75.
* Primary chronic venous insufficiency.
* Patients with known diagnosis of thrombophilia.
* Unavailability of the medical report that documents the prior DVT.
* Post-thrombotic syndrome not confirmed by duplex colour Doppler ultrasound of the lower limbs.
* Solid malignant neoplasm or malignant blood disease in an active state or requiring chemotherapy/radiotherapy.
* Inability to grant consent or refusal to do so.
* Participation in another clinical study in the 4 months prior to screening or during this study.
* Patients who do not comply with the compression therapy required by the protocol 3 (Detailed note after the inclusion criteria).
* Patients with history of hypersensitivity to sulodexide or to any of the excipients of the investigational product.
* Diagnosis of inflammatory joint disease or advanced collagen diseases.
* Pregnancy, breast-feeding or desire to become pregnant during the study.
* Concomitant treatment with anticoagulants, corticosteroids or immunosuppressants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the evolution (change at end of study visit from Baseline ) in the quality of life (QoL). | Participants will be followed for the duration of their study participation, an expected average of 7 months. Change at end of study visit from baseline.
  QOL will be measured using both, the VEINES-QOL and SF-36 questionnaires.
  The total score of the quality-of-life questionnaires will be analysed and the changes that are observed during the study will be expressed as a mean (or median if necessary) with a 95% confidence interval (in the case of the median, using the bootstrapping procedure) and will be analysed to determine the probability of change against the null hypothesis (0 or no change) using a 95% confidence interval for the mean (or the median) and analysis of variance (if the distribution is normal) taking into account the presence of confounding factors.
  Questionnaires will be completed at each study visit:
  V1 "screening" V2 "inclusion" (1 month after screening) V3 (1 month after inclusion) V4 (3 months after inclusion) V5 (6 months after inclusion).

SECONDARY OUTCOMES:
Size of the changes in the axes of the QoL questionnaires. | Participants will be followed for the duration of their study participation, an expected average of 7 months.
  QOL will be measured using both, the VEINES-QOL and SF-36 questionnaires.
  The individual axes of the quality-of-life questionnaires will be analysed in the same way as the total score.
  Questionnaires will be completed at each study visit:
  V1 "screening" V2 "inclusion" (1 month after screening) V3 (1 month after inclusion) V4 (3 months after inclusion) V5 (6 months after inclusion).
Assessment of the degree of correlation between the two QoL questionnaires. | Participants will be followed for the duration of their study participation, an expected average of 7 months.
  QOL will be measured using both, the VEINES-QOL and SF-36 questionnaires.
  The correlation between the total scores on the two questionnaires, if applicable, will be analysed at all times by the Pearson correlation coefficient if both have a normal distribution; otherwise, Spearman's correlation analysis will be used.
  Questionnaires will be completed at each study visit:
  V1 "screening" V2 "inclusion" (1 month after screening) V3 (1 month after inclusion) V4 (3 months after inclusion) V5 (6 months after inclusion).
Extent of the changes and evolution over time of the symptoms/signs evaluated with the VCSS scale (Venous Clinical Severity Score). | Participants will be followed for the duration of their study participation, an expected average of 7 months.
  The changes on the VCSS scale will be reported and analysed in the same way as the primary endpoint
  Questionnaires will be completed at each study visit:
  V1 "screening" V2 "inclusion" (1 month after screening) V3 (1 month after inclusion) V4 (3 months after inclusion) V5 (6 months after inclusion).
Number and percentage by organ and system of Adverse Event. | Participants will be followed for the duration of their study participation, an expected average of 7 months.
  Adverse events will be tabulated and recorded by number and percentage by organ and system. Furthermore, the number of patients with at least one AE, with at least one AE potentially related to the treatment (therefore excluding only those events undoubtedly not related to the treatment), with at least one AE requiring treatment suspension and with at least one serious AE will be tabulated by number and percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Marinel.lo, Study Chair — Hospital de Mataró, Consorci Sanitari del Maresme; Jesús Alós, Principal Investigator — Hospital de Mataró, Consorci Sanitari del Maresme
Locations (17):
- Spain (17):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Espirit Sant de Santa Coloma, Santa Coloma de Gramanet, Barcelona
  - Complejo Hospitalario Universitario de Albacete, Albacete, Castille-La Mancha
  - Hospital Delfos, Barcelona, Catalonia
  - Hospital Universitario de Bellvitge, Barcelona, Catalonia
  - Hospital de Mataró, Mataró (Barcelona), Catalonia
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Catalonia
  - Hospital Universitario HM Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital General de Castellón, Castellon, Valencia
  - Hospital Clínica Platón, Barcelona
  - Hospital Central de la Cruz Roja San José y Santa Adela, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital de Molina, Murcia
  - Hospital Universitari i Politecnic La Fe, Valencia